CLINICAL TRIAL: NCT04558801
Title: The Effects of a Mobile Application-based Lifestyle Counselling on Body Weight Loss in Obese Subjects
Brief Title: Effects of Mobile Application-based Lifestyle Counselling on Body Weight Loss in Obese Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Responsible Party: Principal Investigator, Janne Hukkanen, Professor of Internal Medicine, University of Oulu
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: FeelGood
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mobile application-based lifestyle change program (Experimental): This arm receives the mobile application-based lifestyle change program at baseline. The mobile application-based lifestyle change program consists of twice a week content for the first 6 months, continuing with less frequent content for the following 6 months. The follow-up period is 6 months. Weight is measured and blood samples (lipids, glucose and metabolic syndrome measures) are collected at 0, 6, 12, and 18 months.
  The mobile application-based counselling contains aspects of cognitive behavior therapy and persuasive system design and consists of twice a week reminders, tasks, self-monitoring, and reflection.
  Interventions: Device: Mobile application-based lifestyle change program
- The "waiting-list" control (Active Comparator): The "waiting-list" control arm will receive mobile application-based lifestyle change program after 6 months, following same principles as "Mobile application-based lifestyle change program"-arm, excluding follow-up period (6 months of "waiting list", 6 months of more intense and 6 months of less intense application use).
  Interventions: Device: Mobile application-based lifestyle change program

INTERVENTIONS:
Device: Mobile application-based lifestyle change program — Usage of the Mobile application-based lifestyle change program

SUMMARY:
The aim of the trial is to study the effect of a mobile application-based lifestyle change program on body weight loss in adult subjects with obesity. The main focus is to motivate and support beneficial lifestyle changes targeting long-term weight management.

This study comprises two randomly assigned study arms: mobile application-based lifestyle change program and "waiting-list" control. The mobile application-based lifestyle change program consists of twice a week content for the first 6 months, continuing with less frequent contents for the following 6 months (the length of intervention 12 months). The "waiting-list" control group will receive mobile application-based lifestyle change program after 6 months followed by intervention for 12 months. The main aim is to demonstrate that the users of mobile application-based lifestyle change program lose more weight than controls at 6 month timepoint and weight loss is maintained for 18 months (6 months after the end of mobile application-based lifestyle change program use). Weight is measured and blood samples (lipids, glucose and metabolic syndrome measures) are collected at 0, 6, 12, and 18 months.

The mobile application-based counselling contains aspects of cognitive behavior therapy and persuasive system design and consists of twice a week reminders, tasks, self-monitoring, and reflection.

The main outcome is the decrease in body weight. Secondary outcomes are changes in eating behavior, psychological factors, components of metabolic syndrome (waist circumference, plasma lipid and glucose values, blood pressure), and calculated scores of metabolic condition and adiposity.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index 30 to 40 kg/m2
* Ownership of a smartphone

Exclusion Criteria:

* Untreated hypothyroidism
* Oral glucocorticoid treatment
* Pregnancy or lactation
* No possibility to use mobile phone or tablet
* No knowledge of Finnish language
* Presumed lack of adherence to the study
* Participation in another ongoing weight management program
* Diagnosed or suspicion of cardiovascular disease causing restrictions to exercising
* Bariatric operation planned
* Usage of any anti-obesity drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2020-10-12 (Actual); Primary Completion 2021-07-09 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change in body weight | Baseline to 6 months

SECONDARY OUTCOMES:
Change in body weight | Baseline to 12 months
Change in body weight | Baseline to 18 months
Change in eating behavior | Baseline to 6 months
Change in waist circumference | Baseline to 6 months
Change in blood pressure | Baseline to 6 months
Change in metabolic syndrome status | Baseline to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Janne Hukkanen, MD, PhD, Principal Investigator — University of Oulu, Oulu University Hospital
Locations (1):
- Oulu University Hospital, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No